CLINICAL TRIAL: NCT05708209
Title: The Long Non Coding MALAT1 as a Potential Salivary Diagnostic Biomarker in Oral Squamous Cell Carcinoma Through Targeting mi RNA 124
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Rania Hassan Shalby, Lecturer of Oral Medicine, Fayoum University
Other Study IDs: 19038219038211012
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Long non coding RNA, Oral squamous cell carcinoma, Micro RNA, Salivary biomarkers, MALAT1, Oral cancer biomarkers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: 20 patients with a diagnosis suggestive of OSCC
- Group B: 20 age-and-sex-matched healthy individuals, as normal controls.

SUMMARY:
Objective: is to determine the diagnostic accuracy of lncRNA MALAT1 as a potential salivary biomarker of OSCC as well as assessment of the salivary expression level of miRNA 124 which is targeted by MALAT1. Materials and Methods: Saliva Samples were collected for the quantitative determination of salivary "MALAT1 and mi RNA -124" using quantitative Real-time Polymerase Chain Reaction technique for the two study groups, Group A: 20 patients with a diagnosis suggestive of OSCC and Group B: 20 age-and-sex-matched healthy individuals, as normal controls.

DETAILED DESCRIPTION:
Materials and Methods: Saliva Samples were collected for the quantitative determination of salivary "MALAT1 and mi RNA -124" using quantitative Real-time Polymerase Chain Reaction technique for the two study groups, Group A: 20 patients with a diagnosis suggestive of OSCC and Group B: 20 age-and-sex-matched healthy individuals, as normal controls.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients with OSCC and healthy controls of both sexes.

Exclusion Criteria:

* Patients having systemic diseases such as; liver diseases, cardiovascular disease, nervous system, pulmonary, renal, endocrine, gastrointestinal disorders, or other types of cancer were excluded.

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of oral squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
quantitative determination of salivary non-coding RNAs "MALAT1 | 2 months
  quantitative determination of salivary non-coding RNAs "MALAT1 using quantitative Real-time Polymerase Chain Reaction technique (qRT-PCR) in the whole unstimulated saliva

SECONDARY OUTCOMES:
quantitative determination of salivary mi RNA -124" | 2 months
  quantitative determination of salivary mi RNA -124" using quantitative Real-time Polymerase Chain Reaction technique (qRT-PCR) in the whole unstimulated saliva

CONTACTS AND LOCATIONS:
Locations (1):
- Rania Hassan Shalby, Giza, Egypt